CLINICAL TRIAL: NCT04654611
Title: Ocular Surface Conditions in Asian Glaucoma Patients With Existing Corneal Disorders Switching From Preserved Prostaglandin Analogues Monotherapy to Preservative-free Tafluprost
Brief Title: Tafluprost Preservative Free Switch Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tun Hussein Onn National Eye Hospital (Other)
Responsible Party: Principal Investigator, Thanendthire Sangapillai, Principal Investigator, Ophthalmology Senior Registrar, Tun Hussein Onn National Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-11-23; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Other): The intervention will be preservative free tafluprost 0.0015% topical ophthalmic solution given once daily for the study duration.
  Interventions: Drug: preservative free tafluprost 0.0015%

INTERVENTIONS:
Drug: preservative free tafluprost 0.0015% — preservative free prostaglandin analogue option for treatment of primary open angle glaucoma and ocular hypertension patients

SUMMARY:
This study is conducted to document the effect of switching from preserved prostaglandin analogues monotherapy to preservative free tafluprost 0.0015%. The endpoints analyzed are side effect improvement in these patients.

DETAILED DESCRIPTION:
Importance: Glaucoma medications are often preserved with agents such as benzalkonium chloride, which commonly lead to ocular surface diseases.

Background: To investigate the effect of switching to a preservative-free prostaglandin analogue, tafluprost 0.0015% on treatment tolerability and ocular surface diseases.

Design: This was a prospective, open label, non-randomised, observational study performed in a single hospital.

Participants: Patients of Asian descent who have primary open angle glaucoma and ocular hypertension (n = 28), who received preserved prostaglandin monotherapy for longer than 3 months, and has a National Eye Institute ocular surface staining scale score higher than 1.

Methods: Patients were switched from preserved prostaglandin monotherapy to preservative-free tafluprost 0.0015%. Patients were analysed at baseline (Visit 0), 1 month (Visit 1) and 3 months (Visit 2).

Main Outcome Measures: The main parameter measured is the change in the fluorescein staining score at Visit 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 21 years or older and those who can provide informed consent.
2. Patients who have corneal disorders due to the prostaglandin usage. (At least one eye must have a score above 1 on the NEI scale)
3. Intraocular pressure (IOP) ≤ 21 mm Hg in the study eye at the screening examination (under treatment)
4. If only one eye is eligible, it is to be evaluated. If both eyes are eligible, then the eye with a higher NEI score will be selected for evaluation.
5. Pretreatment must be monotherapy with any of the following preserved ophthalmic solutions; latanoprost, travoprost, bimatoprost or tafluprost and its period must be longer than 3 months.
6. Outpatients who can visit the clinic on the designated day as instructed by the physician.
7. A best-corrected ETDRS visual acuity score of +0.6 logMAR (Snellen equivalent of 20 ⁄ 80) or better in each eye.

Exclusion Criteria:

1. Those with severe visual field disorder (Mean deviation of 15 dB or worse)
2. Those with a history of ocular surgeries (such as corneal refractive surgery, intraocular surgery including ocular laser treatment which may affect the patient's ocular surface condition) within 6 months prior to the study initiation.
3. Those with severe dry eye (those in need of drug to treat dry eye), ocular allergy, ocular infection or ocular inflammation
4. Those who need to use systemic or ophthalmic steroids (excluding topical skin steroidal ointment) and anti-glaucoma agents other than latanoprost, travoprost, bimatoprost or preservative free tafluprost ophthalmic solution
5. Female patients who are pregnant, nursing or lactating
6. Those with a history of drug allergy (hypersensitivity) to the drugs to be used during the study period (anesthetic ophthalmic solution, fluorescein, etc.) or similar drugs to the investigational product
7. Those who need to wear contact lenses during the study period
8. Any corneal abnormality or other condition preventing reliable applanation tonometry
9. Anterior chamber angle less than grade 2 according to Schaffer classification as measured by Gonioscopy
10. Any uncontrolled systemic disease (e.g. hypertension, diabetes)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in the fluorescein staining score (NEI) at Visit 2 | 3 months
  The fluorescein stained area of the cornea will be measured according to the National Eye Institute/Industry (NEI/I) method. NEI grading scale consists of a grid that divides the corneal area into five sections, each of which is assigned a score between zero and 3 depending of the amount and distribution of Corneal Fluorescein Stain (CFS); the total CFS score ranges from 0/15 (absence of corneal epitheliopathy) to 15/15 (severe epitheliopathy)

CONTACTS AND LOCATIONS:
Overall Officials: Hsien Han Lim, Principal Investigator — Tun Hussein Onn National Eye Hospital
Locations (1):
- THONEH, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No